CLINICAL TRIAL: NCT05901766
Title: Effect of Maternal Supplementation With an Iodine-containing Multiple Micronutrient During Lactation on Infant Iodine Status, Thyroid Function and Neurodevelopment
Brief Title: Effect of Iodine-containing Multiple Micronutrient During Lactation on Infant Neurodevelopment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Addis Continental Institute of Public Health (Other); Brigham and Women's Hospital (Other); Johns Hopkins Bloomberg School of Public Health (Other); University of South Carolina (Other)
Responsible Party: Principal Investigator, Anne Shee CC Lee, Levinger Family Professor of Pediatrics, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002634
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Iodine Deficiency; Nutrition Poor; Development, Infant; Breastfeeding
MeSH Terms: conditions — Malnutrition; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Individually randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iodine Containing Multiple Micronutrient (UNIMAP) (Experimental): UNIMAP 1 tablet po once daily from birth to 6 months postpartum
  Interventions: Dietary Supplement: UNIMAP Multiple Micronutrient Supplement
- Routine postnatal care (No Intervention): Routine postnatal care per Ethiopian Ministry of Health guidelines

INTERVENTIONS:
Dietary Supplement: UNIMAP Multiple Micronutrient Supplement — Iodine Containing Multiple Micronutrient Supplement once daily
  Arms: Iodine Containing Multiple Micronutrient (UNIMAP)

SUMMARY:
The goal of this clinical trial is to learn about the effects of iodine-containing multiple micronutrient supplements provided to breastfeeding mothers who live in settings with mild iodine deficiency.

The main questions it aims to answer are:

1. What are the effects of iodine-containing multiple micronutrient supplements provided to breastfeeding mothers on infant development, as measured by electroencephalography/visual evoked potentials?
2. What are the effects of iodine-containing multiple micronutrient supplements on breast milk concentrations of iodine, and infant iodine and thyroid status?
3. How do iodine and iron interact with each other to affect thyroid function in the mother during lactation?

Participants will be randomized to receive a daily multiple micronutrient tablet containing iodine (UNIMAPP) for 6 months postpartum, or routine postnatal care per Ethiopia Ministry of Health. Mothers will provide a breast milk sample and blood at 3 and 6 months postpartum. Infants will provide a urine sample and drop of blood, and have a neurodevelopmental assessment at 3 and 6 months.

Researchers will compare the groups that received the iodine-containing micronutrient supplement with the group that received routine care and see if there were any benefits on infant development and iodine and thyroid status in the mother and baby.

ELIGIBILITY:
Inclusion Criteria:

* Intention to breast feed at least 3 months
* Birth weight >2000g

Exclusion Criteria:

* Intention to primarily feed by alternative sources (formula, animal milk)
* Multiple pregnancy
* Infant with major congenital anomalies
* Infants with severe morbidity or developmental disorder
* Mother with HIV or chronic renal disease
* Plan to move out of study catchment area
* Does not agree to follow up or EEG/VEP

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual Evoked Potentials | 6 months post partum
  P1 Latency
BMIC | 1 month post partum
  Breast Milk Iodine Concentration at 1 month

SECONDARY OUTCOMES:
EEG Fc | 6 months
  EEG Functional Connectivity
Infant HCAZ at 6 months | 6 months
  Infant head circumference Z-score
Infant UIC | 6 months
  Infant Urine Iodine Concentration
Infant Tg | 6 months
  Dried blood spot thyroglobulin
Infant TSH | 6 months
  Thyroid Stimulating Hormone

IPD SHARING:
Plan to Share IPD: Undecided